CLINICAL TRIAL: NCT01375738
Title: The Effect and Mechanism of Improving Diabetes by Reconstruction Methods in Gastric Cancer Patients With DM Who Receive Surgical Treatment
Brief Title: Improving Diabetes by Reconstruction Methods in Gastric Cancer Patients With Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, ji yeong an, assistant professor, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2011-0109
Record Dates: First submitted 2011-05-27; First posted 2011-06-17 (Estimated); Last update posted 2012-09-13 (Estimated); Status verified 2012-09

CONDITIONS: Gastric Cancer; Diabetes
Keywords: Early gastric cancer
MeSH Terms: conditions — Stomach Neoplasms; Diabetes Mellitus | interventions — Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gastroduodenostomy (Active Comparator): Arm 1: undergo gastroduodenostomy after distal gastrectomy for gastric cancer
  Interventions: Procedure: Gastroduodenostomy
- Roux-en Y gastrojejunostomy (Experimental): Arm 2: undergo Roux-en Y gastrojejunostomy after distal gastrectomy for gastric cancer
  Interventions: Procedure: Roux-en Y gastrojejunostomy

INTERVENTIONS:
Procedure: Roux-en Y gastrojejunostomy — After subtotal gastrectomy with lymph node dissection, the jejunum is transected 25~30cm distal to the ligament of Treitz. Distal jejunum is drawn up and sutured to the gastric remnant and the proximal jejunum is anastomosed to the distal jejunum at 30~40cm from the new gastric-jejunal junction.
  Arms: Roux-en Y gastrojejunostomy
Procedure: Gastroduodenostomy — After subtotal gastrectomy with lymph node dissection, the gastric remnant is anastomosed to duodenum 1st portion with circular or linear staplers and the artificial lesser curvature is repaired with linear stapler.
  Arms: Gastroduodenostomy

SUMMARY:
This study is to investigate the effect of gastrectomy on remission of type 2 diabetes in patients with gastric cancer and type 2 diabetes, to investigate the mechanism of blood glucose alteration and intestinal hormonal signaling by the reconstruction methods, and to evaluate the applicability and efficacy of Roux-en-Y gastrojejunostomy after gastrectomy in gastric cancer patients with diabetes.

DETAILED DESCRIPTION:
Purpose:

* To investigate the effect of gastrectomy on remission of type 2 diabetes in patients with gastric cancer and type 2 diabetes
* To investigate the mechanism of blood glucose alteration and intestinal hormonal signaling by the reconstruction methods
* To evaluate the applicability and efficacy of Roux-en-Y gastrojejunostomy after gastrectomy in gastric cancer patients with diabetes

Contents:

* Evaluation of the status of diabetes in gastric cancer patients with DM after gastrectomy

  * Comparison of two reconstruction types after gastrectomy Bypass duodenum and upper jejunum: Roux-en-Y gastrojejunostomy Preservation of duodenal passage: Gastroduodenostomy
  * Analysis for biochemical markers reflecting diabetic status: fasting glucose, postprandial 2h glucose, HbA1c, C-peptide, lipid profile
* Correlation of parameters associated with diabetes and GI hormones

  * Measurement of GI hormones which have an effect on glucose tolerance

    * Insulin, glucagon, IGF-1, GLP-1, Neuropeptide Y, Ghrelin, Leptin
  * Correlation of reconstruction methods, parameters of diabetes and GI hormone levels
  * Evaluation of mechanism of Roux-en-Y gastrojejunostomy on controlling diabetes
* Evaluation of Feasibility of Roux-en-Y gastrojejunostomy in gastric cancer surgery in patients with DM

  * Degree of high blood glucose control, the amount of antidiabetic medication, costs for DM treatment, quality of life assessment
  * Analysis for the mechanism of gastrointestinal physiology to diabetes control

ELIGIBILITY:
Inclusion Criteria:

* Patient who are older than 20 years and younger than 80 years
* Histologically confirmed gastric adenocarcinoma located lower one third of stomach
* Postoperative confirmed pT1N0, pT2N0, pT1N1
* Informed consent

Exclusion Criteria:

* Previous history of treatment for other malignancy or inflammatory disease
* Preoperative uncontrolled serious comorbidity
* Vulnerable Subjects(pregnant women, children, cognitively impaired persons etc.)
* Patient who experience any complications requiring reoperation following gastrectomy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-07; Primary Completion 2013-06 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Blood sugar stabilization after gastrectomy | three months after surgery
  By comparing the difference between fasting blood sugar and postprandial blood glucose, blood sugar stabilization after gastrectomy will be maesured.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

REFERENCES:
- [Background] Yang J, Li C, Liu H, Gu H, Chen P, Liu B. Effects of subtotal gastrectomy and Roux-en-Y gastrojejunostomy on the clinical outcome of type 2 diabetes mellitus. J Surg Res. 2010 Nov;164(1):e67-71. doi: 10.1016/j.jss.2010.07.004. Epub 2010 Jul 30. PMID 20863527
- [Derived] Nishizaki D, Ganeko R, Hoshino N, Hida K, Obama K, Furukawa TA, Sakai Y, Watanabe N. Roux-en-Y versus Billroth-I reconstruction after distal gastrectomy for gastric cancer. Cochrane Database Syst Rev. 2021 Sep 15;9(9):CD012998. doi: 10.1002/14651858.CD012998.pub2. PMID 34523717